CLINICAL TRIAL: NCT06403397
Title: Assessing the Impact of Monitor Maintenance Package Utilization on Patient Monitor Alarms and Nurse Alarm Fatigue
Brief Title: Assessing the Impact of Monitor Maintenance Package Utilization
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Istanbul Demiroglu Bilim University (Other)
Responsible Party: Principal Investigator, Ogretim Uyesi Serpil Topcu, Assistant Professor, Istanbul Demiroglu Bilim University
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: Remember Me Tool
Record Dates: First submitted 2024-04-29; First posted 2024-05-07 (Actual); Last update posted 2024-05-07 (Actual); Status verified 2024-05

CONDITIONS: Alarm Fatigue; Patient Safety
Keywords: alarm fatigue; Intensive care unit; Nurse-driven monitoring bundle; patient safety
MeSH Terms: conditions — Alert Fatigue, Health Personnel

STUDY DESIGN:
Intervention Model Description: This study is a cross-controlled experimental research conducted to determine the effect of using the CEASE care package on patient monitor alarms and nurse alarm fatigue in adult intensive care units
Who Masked: Care Provider
Masking Description: The population of the study consists of all nurses working in the intensive care units of Prof. Dr. Cemil Taşcıoğlu City Hospital. There are a total of 142 nurses working in the adult intensive care units of the hospital.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental group (Experimental): * Working in the intensive care unit,
  * Willing to participate in the study voluntarily,
  * Nurses willing to use the monitor alarm control tool.
  Interventions: Other: Experimental group: CEASE Care Package and Remember Me Tool
- Control group (No Intervention): * Working in the intensive care unit,
  * Willing to participate in the study voluntarily,

INTERVENTIONS:
Other: Experimental group: CEASE Care Package and Remember Me Tool — Before the intervention, the intervention group will first undergo the 'Nurse Identification Form' and the 'Alarm Fatigue Scale'. The current root cause analysis of monitor alarms in the clinical setting will be conducted through the 'CEASE Care Package' and the 'Current Situation Analysis Form'. Each patient monitor in the intensive care unit will be observed and recorded by two observers for a period of 24 hours.The Monitor Alarm Control Tool - "Remember Me" will be attached beneath each monitor to facilitate easier monitoring by nurses. Nurses are expected to use the tool for a period of 15 days. After intervention; Two observers will conduct a re-evaluation using the "CEASE Care Package" and the "Current Status Analysis Form". Monitor alarms will be continuously assessed and recorded for 24 hours. Following the completion of this stage, the "Alarm Fatigue Scale" will be reapplied to the intervention group.
  Arms: Experimental group

SUMMARY:
Bedside monitors are frequently used in monitoring vital signs of critically ill patients. Nurses working in healthcare facilities, especially in intensive care units, are required to manage devices with different alarm threshold values, categories, and types of alerts, leading to alarm fatigue. In response to this serious threat to patient safety, the FDA and The Joint Commission worked to develop strategies to address alarm fatigue in 2011. Alarm monitoring, identification of the cause, and silencing are typically performed by nurses. When reviewing alarm control studies in the literature, the CEASE care package developed by Levis et al. in 2019 was encountered. The tool was developed for personalized clinical alarm monitoring for the patient.

DETAILED DESCRIPTION:
Bedside monitors are frequently used in monitoring vital signs of critically ill patients. Patient monitors assist healthcare professionals in continuous monitoring of basic vital signs such as EKG (electrocardiogram), blood pressure, pulse oximetry, respiration, as well as advanced hemodynamic parameters like central venous pressure, pulmonary artery pressure. These devices alert healthcare personnel visually and audibly in case of any abnormality in the monitored parameters. According to the Sentinel Event Alert report published by The Joint Commission (TJC) in 2013, each unit can receive thousands of alarm alerts in a single day. It is stated that 85% to 99% of these alarms are either not related to the patient's clinical condition, false, or do not require any action. This situation leads to necessary alarms being silenced, ignored, or muted, thereby threatening patient safety. Thousands of patient injuries and deaths have been reported due to alarm system errors. The main reasons for alarm errors include failure to recognize the alarm, desensitization in nurses, inadequate training in monitor usage, decreased response time to alarms, deficiencies in device interface design, equipment failures, and staff shortages. Monitor alarms occur in a hierarchy of high, medium, and low priority. Each hierarchical alarm produces a different auditory tone. Clinicians use these alarm tones to determine the urgency level and appropriate alarm response. When clinically irrelevant alarms occur more frequently, there is a higher likelihood of overall alarm fatigue. Nurses working in healthcare facilities, especially in intensive care units, are required to manage devices with different alarm threshold values, categories, and types of alerts, leading to alarm fatigue. Alarm fatigue is defined as healthcare workers becoming desensitized and indifferent to many recurring or simultaneous alarm sounds. In response to this serious threat to patient safety, the FDA and The Joint Commission worked to develop strategies to address alarm fatigue in 2011. The published report emphasizes the need to identify the problem clinically and develop solution strategies tailored to the problem, to be implemented alongside general standard interventions. The report primarily focuses on adjusting alarm parameters appropriately and establishing clinic-specific protocols and procedures. Alarm monitoring, identification of the cause, and silencing are typically performed by nurses. When reviewing alarm control studies in the literature, the CEASE care package developed by Levis et al. in 2019 was encountered. The tool was developed for personalized clinical alarm monitoring for the patient. The name CEASE is formed by combining the initials of the words Communication, Electrodes, Appropriateness, Setup, and Education. Researchers found a decrease in the number of monitor alarms and alarm fatigue levels in nurses after using the CEASE care package. More supportive studies are needed for the widespread adoption of this package in clinics. In this study, the investigators aimed to demonstrate a reduction in unnecessary alarm counts and a decrease in nurse alarm fatigue levels with the use of the CEASE care package.

ELIGIBILITY:
Inclusion Criteria:

* Working in the intensive care unit,
* Willing to participate in the study voluntarily,
* Nurses willing to use the monitor alarm control tool (for intervention group).

Exclusion Criteria:

* Nurses who leave the intensive care unit during the data collection process and those who do not use the monitor alarm control tool

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 142 (Estimated)
Dates: Start 2024-06-15 (Estimated); Primary Completion 2024-08-15 (Estimated); Study Completion 2024-12-15 (Estimated)

PRIMARY OUTCOMES:
The use of the CEASE care package tool will result in a decrease in the number of alarms in the intensive care unit end of the 3 weeks. | 2 months
  This outcome will measured by Current Situation Analysis Form and CEASE care package tool.
The use of the CEASE care package tool will lead to a reduction in alarm fatigue levels end of the 3 weeks. | 2 months
  This outcome will measured by alarm fatigue scale.

CONTACTS AND LOCATIONS:
Locations (1):
- Demiroğlu Bilim University, Istanbul, Şişli, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
Researchers may share IPD data after the completion and publication of the study.

REFERENCES:
- [Background] Schmid F, Goepfert MS, Reuter DA. Patient monitoring alarms in the ICU and in the operating room. Crit Care. 2013 Mar 19;17(2):216. doi: 10.1186/cc12525. No abstract available. PMID 23510435
- [Background] Joint Commission. Medical device alarm safety in hospitals. Sentinel Event Alert. 2013 Apr 8;(50):1-3. No abstract available. PMID 23767076
- [Background] De Vaux L, Cooper D, Knudson K, Gasperini M, Rodgerson K, Funk M. Reduction of Nonactionable Alarms in Medical Intensive Care. Biomed Instrum Technol. 2017 Feb;51(s2):58-61. doi: 10.2345/0899-8205-51.s2.58. No abstract available. PMID 28296452
- [Background] Clark, T., David, Y., & Baretich, M. Impact of clinical alarms on patient safety. ACCE Healthcare Technology Foundation 2006: 1-20
- [Background] Sendelbach S, Funk M. Alarm fatigue: a patient safety concern. AACN Adv Crit Care. 2013 Oct-Dec;24(4):378-86; quiz 387-8. doi: 10.1097/NCI.0b013e3182a903f9. PMID 24153215
- [Background] Graham KC, Cvach M. Monitor alarm fatigue: standardizing use of physiological monitors and decreasing nuisance alarms. Am J Crit Care. 2010 Jan;19(1):28-34; quiz 35. doi: 10.4037/ajcc2010651. PMID 20045845
- [Background] Association for the Advancement of Medical Instrumentation (2011). A siren call to action: Priority issues from the medical device alarms summit. Clinical Alarms AAMI Summit Proceedings, 5(6).
- [Background] Cvach M. Monitor alarm fatigue: an integrative review. Biomed Instrum Technol. 2012 Jul-Aug;46(4):268-77. doi: 10.2345/0899-8205-46.4.268. PMID 22839984
- [Background] Erbay-Dalli O, Bagci-Derinpinar K. Adaptation and validation of the Turkish version of the alarm fatigue assessment questionnaire. Enferm Intensiva (Engl Ed). 2024 Apr-Jun;35(2):114-123. doi: 10.1016/j.enfie.2023.09.001. Epub 2023 Oct 5. PMID 37805362
- [Background] Alarm management. Crit Care Nurse. 2013 Oct;33(5):83-6. No abstract available. PMID 24085833
- [Background] Ashrafi, S., Najafi Mehri, S., & Nehrir, B. (2017). Designing an Alarm Fatigue Assessment Questionnaire: Evaluation of the Validity and Reliability of an Instrument. Journal of Critical Care Nursing, 10(4), 0-0.
- [Background] Lewis CL, Oster CA. Research Outcomes of Implementing CEASE: An Innovative, Nurse-Driven, Evidence-Based, Patient-Customized Monitoring Bundle to Decrease Alarm Fatigue in the Intensive Care Unit/Step-down Unit. Dimens Crit Care Nurs. 2019 May/Jun;38(3):160-173. doi: 10.1097/DCC.0000000000000357. PMID 30946125